CLINICAL TRIAL: NCT00545103
Title: A Phase III, Randomised, Double-Blind, Dose-Response, Stratified, Placebo-Controlled Study Evaluating the Safety and Efficacy of SPD476 Versus Placebo Over 104 Weeks in the Prevention of Recurrence of Diverticulitis.
Brief Title: Prevention of Recurrence of Diverticulitis
Acronym: PREVENT2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: SPD476-314; 2007-004896-20 (EudraCT Number)
Record Dates: First submitted 2007-10-16; First posted 2007-10-17 (Estimated); Results first posted 2012-12-19 (Estimated); Last update posted 2021-06-11 (Actual); Status verified 2021-05

CONDITIONS: Diverticulitis
MeSH Terms: conditions — Diverticulitis | interventions — Mesalamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- SPD476 (1.2 g) (Experimental)
  Interventions: Drug: SPD476, MMX™ mesalazine, 1.2g extended release tablet
- SPD476 (2.4 g) (Experimental)
  Interventions: Drug: SPD476, MMX™ mesalazine, 2.4g extended release tablet
- SPD476 (4.8 g) (Experimental)
  Interventions: Drug: SPD476, MMX™ mesalazine, 4.8g extended release tablet
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SPD476, MMX™ mesalazine, 1.2g extended release tablet — SPD476 1.2g administered Once Daily (QD)
  Other Names: LIALDA
  Arms: SPD476 (1.2 g)
Drug: SPD476, MMX™ mesalazine, 2.4g extended release tablet — SPD476 2.4g administered Once Daily (QD)
  Other Names: LIALDA
  Arms: SPD476 (2.4 g)
Drug: SPD476, MMX™ mesalazine, 4.8g extended release tablet — SPD476 4.8g administered Once Daily (QD)
  Other Names: LIALDA
  Arms: SPD476 (4.8 g)
Drug: Placebo — Placebo administered Once Daily (QD)
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether SPD476 is effective in reducing recurrence of diverticulitis.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females =>18yrs of age.
2. If female of childbearing potential (FOCP), has demonstrated a negative beta HCG (human chorionic gonadotropin) serum pregnancy test, and agrees to comply with any applicable contraceptive requirements of the protocol
3. An episode of acute diverticulitis that resolved without colonic resection.
4. Confirmation of diverticulosis via endoscopic evaluation of the sigmoid colon with at least three diverticula noted

Exclusion Criteria:

1. Previous colorectal surgery, including surgical intervention for diverticular disease (with the exception of haemorrhoidectomy, colonic removal of polyps, and appendectomy)
2. Active peptic ulcer disease
3. History of or current presence of inflammatory bowel disease (IBD)
4. Subjects with active irritable bowel syndrome (IBS) requiring ongoing medication
5. Allergy or hypersensitivity to aspirin or related compounds
6. Allergy to radiologic contrast agents
7. Use of another Investigational product within 30 days of Baseline
8. Use of antibiotic therapy within 4 weeks of Baseline
9. Within 14 days of Baseline, use of prebiotic, probiotic or 5-ASA medications, as well as drugs active at the 5HT-receptor or anti-spasmodic agents
10. Use of systemic or rectal steroids within 6 weeks of Baseline. Use of inhaled or nasal steroids is acceptable
11. Use of anti-inflammatory drugs, (NSIADs, COX-2 inhibitors) including aspirin (except for cardiac prophylaxis) and ibuprofen, on a regular and ongoing basis
12. History of alcohol or other substance abuse within the previous year
13. Active or recent history of endometriosis or dysmenorrhoea within 6 months prior to Baseline
14. Females who are lactating

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 592 (Actual)
Dates: Start 2007-12-06 (Actual); Primary Completion 2011-11-28 (Actual); Study Completion 2011-11-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (131):
- United States (59):
  - Birmingham Gastroenterology Associates, PC, Birmingham, Alabama
  - Alabama Clinical Therapeutics, LLC, Birmingham, Alabama
  - Medical Affiliated Research Center, Inc, Huntsville, Alabama
  - Alabama Digestive Disorders Center, PC, Huntsville, Alabama
  - Genova Clinical Research, Tucson, Arizona
  - Digestive and Liver Disease Specialists, Garden Grove, California
  - High Desert Gastroenterology, Inc., Lancaster, California
  - VA Long Beach Healthcare System, Long Beach, California
  - CA Physicians Research Alliance, Oceanside, California
  - Digestive Care Medical Center, San Carlos, California
  - Rider Research Group, San Francisco, California
  - Huntington Medical Foundation, San Marino, California
  - Clinical Research of the Rockies, Lafayette, Colorado
  - Arapahoe Gastroenterology, PC, Littleton, Colorado
  - Litchfield County Gastroenterology Associates, LLC, Torrington, Connecticut
  - Madeleine DuPree, MD, Boynton Beach, Florida
  - Palmetto Research LLC, Hialeah, Florida
  - Mark Lamet, MD, Hollywood, Florida
  - Digestive Disease Consultants, Maitland, Florida
  - University of Miami Miller School of Medicine, Miami, Florida
  - University of Miami, Miami, Florida
  - Miami Research Associates, Miami, Florida
  - United Medical Research, New Smyrna Beach, Florida
  - West Wind'r Research & Development, Tampa, Florida
  - Atlanta Gastroenterology Associates, Marietta, Georgia
  - Gastrointestinal Clinical of Quad Cities, Davenport, Iowa
  - Sunflower Medical Group, Mission, Kansas
  - Kansas Medical Clinic, Topeka, Kansas
  - Gastroenterology Associates, LLC, Baton Rouge, Louisiana
  - Louisiana Research Center, LLC, Shreveport, Louisiana
  - Maryland Clinical Trials, Annapolis, Maryland
  - Chevy Chase Clinical Research, Chevy Chase, Maryland
  - Mid Atlantic Medical Research Centers, Hollywood, Maryland
  - Charm City Research, LLC, Lutherville, Maryland
  - Shah Associates, LLC, Prince Frederick, Maryland
  - Clinical Research Institute of Michigan, LLC, Chesterfield, Michigan
  - Center for Digestive Health, Troy, Michigan
  - Gastrointestinal Associates, PA, Jackson, Mississippi
  - Center for Digestive & Liver Diseases, Inc, Mexico, Missouri
  - Sundance Clinical Research, St Louis, Missouri
  - The Gastroenterology Group of South Jersey, Vineland, New Jersey
  - NY Center for Clinical Research, Lake Success, New York
  - Concorde Medical Group, New York, New York
  - Cumberland Research Associates, Fayetteville, North Carolina
  - LeBauer Research Associates, PA, Greensboro, North Carolina
  - Wake Research Associates, Raleigh, North Carolina
  - Digestive Health Specialists, Winston-Salem, North Carolina
  - Consultants for Clinical Research, Cincinnati, Ohio
  - Digestive Specialists Inc., Dayton, Ohio
  - AMH Feasterville Family Health Care Center, Feasterville, Pennsylvania
  - Digestive Disorders Center, Pittsburgh, Pennsylvania
  - Clinsearch, LLC, Chattanooga, Tennessee
  - Memphis Gastroenterology Group, PC, Germantown, Tennessee
  - Houston Endoscopy and Research Center, Houston, Texas
  - Hidalgo Clinical Research, San Antonio, Texas
  - Physician Research Options, Murray, Utah
  - Granite Peaks Gastroenterology, Sandy City, Utah
  - Northwest Gastroenerology Associates, Bellevue, Washington
  - Seattle Gastroenterology Associates, Seattle, Washington
- Brazil (10):
  - Instituto Goiano de Gastroenterologia e Endoscopia Digestiva Ltda., Goiânia, Goiás
  - Universidade Federal de Juiz de Fora, Juiz de Fora, Minas Gerais
  - Hospital Universitário Clementino Fraga Filho, Rio de Janeiro, Rio de Janeiro
  - Hospital de Clinicas de Porto Alegre, Porto Alegre, Rio Grande do Sul
  - Hospital Sao Lucas PUCRS, Porto Alegre, Rio Grande do Sul
  - Fundacao Universidade Federal do Rio Grande - Hopsital Universitario, Rio Grande, Rio Grande do Sul
  - Unidade Integrada de Gastroenterologia UNIGASTRO, Campinas, São Paulo
  - Irmandade da Santa Casa de Misericordia de Santos, Santos, São Paulo
  - Hospital Universitario Pedro Ernesto, Rio de Janeiro
  - Centro de Pesquisas Clinicas- CPCLIN, São Paulo
- Canada (9):
  - Liver and Intestinal Research Centre, Vancouver, British Columbia
  - Topsail Road Medical Clinic, St. John's, Newfoundland and Labrador
  - Corunna Medical Research Centre, Corunna, Ontario
  - Cleveland Clinic Canada, Toronto, Ontario
  - Hotel-Dieu de Levis, Lévis, Quebec
  - Omnispec Clinical Research, Mirabel, Quebec
  - Hopital Maisonneuve-Rosemont, Montreal, Quebec
  - Gastroenterology Centre, Pointe-Claire, Quebec
  - Q&T Research, Sherbrooke, Quebec
- Finland (5):
  - Suomen Terveystalo Oyj, Jyväskylä
  - Kuopio University Hospital, Kuopio
  - Päijat-Häme Central Hospital, Lahti
  - Oulu University Hospital, Oulu
  - Vaasa Central Hospital, Vaasa
- Germany (9):
  - Synexus ClinPharm GmbH Berlin, Berlin, Berlin (Hellersdorf)
  - Gastrologische Gemeinschaftspraxis Herne im Ärztehaus am Evangelischen Krankenhaus Herne, Herne, Nord-Rhein-Wesfalen
  - Synexus ClinPharm International GmbH, Bochum
  - Synexus ClinPharm International GmbH, Frankfurt
  - Synexus ClinPharm International GmbH, Görlitz
  - Universitätsklinikum Schleswig-Holstein, Kiel
  - Synexus ClinPharm International GmbH, Leipzig
  - Synexus ClinPharm International GmbH, Magdeburg
  - Synexus ClinPharm International GmbH, Potsdam
- Hungary (6):
  - Peterfy Hospital, Dept. Of Gastroenterology, Budapest
  - University of Debrecen, 3rd Dept. Of Medicine, Debrecen
  - Bekes Megyei Kepviselotestulet Pandy Kalman Korhaza, Endoszkopos laboratorium, Gyula
  - Kaposi Mór Teaching Hospital, Kaposvár
  - Karolina Hospital, Dept. of Internal Medicine and Gastroenterology, Mosonmagyaróvár
  - Jávorszky Ödön Városi Kórhaz, II. Belgyógyászat, Vác
- Italy (9):
  - Ospedale Valduce, Como
  - Ospedale Fatebenefratelli ed Oftalmico, Milan
  - Universita degli Studi di Padova, Padua
  - U.O. di Gastroenterologia ed Endoscopia digestiva Torre delle Medicine Azienda Ospedaliera di Parma, Parma
  - Universita di Pavia Cattedra di Gastroenterologia Dipartimento di Medicina, Pavia
  - Azienda Ospedaliera Universitaria Policlinico Tor Vergata, Roma
  - San Camillo Forlanini, Roma
  - Policlinico Univeritario A Gemelli, Roma
  - Policlinico Univeritario A. Gemelli, Roma
- Netherlands (5):
  - Meander Medisch Centrum, Amersfoort
  - VU Medisch Centrum, Amsterdam
  - Academisch Ziekenhuis Maastricht, Maastricht
  - Ikazia Ziekenhuis, Rotterdam
  - St. Jans Gashuis, Weert
- Romania (7):
  - CMI de Gastroenterologie Dobru Daniela, Târgu Mureş, Mureș County
  - Spitalul Clinic "Dr. I. Cantacuzino", Bucharest
  - Institutul Clinic Fundeni, Bucharest
  - Spitalul Universitar de Urgenta Bucuresti, Bucharest
  - Centrul Medical Galenus, Târgu Mureş
  - Cabinet Particular Policlinic Algomed SRL, Timișoara
  - Policlinica "Dr. Citu" SRL, Timișoara
- South Africa (12):
  - Panorama Medi-Clinic, Cape Town, Western Cape
  - Universitas Hospital, Bloemfontein
  - Harold Bloch, Cape Town
  - Panorama Medi-Clinic, Cape Town
  - Louis Leipoldt Medical Centre, Cape Town
  - Kingsbury Hospital, Cape Town
  - Parklands Medical Centre, Durban
  - Chelmsford Medical Centre 2, Durban
  - Milpark Hospital, Johannesburg
  - Linksfield Park Clinic, Johannesburg
  - Johannesburg General Hospital, Johannesburg
  - Kloof Medi-Clinic, Pretoria

REFERENCES:
- [Derived] Raskin JB, Kamm MA, Jamal MM, Marquez J, Melzer E, Schoen RE, Szaloki T, Barrett K, Streck P. Mesalamine did not prevent recurrent diverticulitis in phase 3 controlled trials. Gastroenterology. 2014 Oct;147(4):793-802. doi: 10.1053/j.gastro.2014.07.004. Epub 2014 Jul 16. PMID 25038431

RESULTS

PARTICIPANT FLOW:
Groups:
- SPD476 (1.2 g): 1.2 g administered orally once daily
- SPD476 (2.4 g): 2.4 g administered orally once daily
- SPD476 (4.8 g): 4.8 g administered orally once daily
- Placebo: Placebo administered orally once daily
Period: Overall Study
Arm/Group | SPD476 (1.2 g) | SPD476 (2.4 g) | SPD476 (4.8 g) | Placebo
Started | 148 | 148 | 150 | 146
Completed | 73 | 70 | 74 | 76
Not Completed | 75 | 78 | 76 | 70
Not completed — Lack of Efficacy | 48 | 45 | 31 | 27
Not completed — Withdrawal by Subject | 6 | 10 | 18 | 22
Not completed — Adverse Event | 11 | 12 | 17 | 10
Not completed — Lost to Follow-up | 4 | 6 | 3 | 4
Not completed — Protocol Violation | 1 | 2 | 3 | 0
Not completed — Suspected recurrence of diverticulitis | 1 | 0 | 0 | 3
Not completed — Difficult to open package | 0 | 0 | 0 | 1
Not completed — Investigational product not taken | 1 | 0 | 0 | 1
Not completed — Wish to start a family | 0 | 0 | 0 | 1
Not completed — Diverticulitis crisis | 0 | 0 | 0 | 1
Not completed — Personal reasons | 1 | 0 | 0 | 0
Not completed — Subject's decision | 1 | 0 | 0 | 0
Not completed — Noncompliance | 0 | 1 | 0 | 0
Not completed — Investigator decision | 0 | 0 | 1 | 0
Not completed — Subject moved | 0 | 1 | 0 | 0
Not completed — Use of prohibited medication | 0 | 0 | 1 | 0
Not completed — Does not want to take study drug anymore | 1 | 0 | 1 | 0
Not completed — Subject met endpoint under protocol v. 1 | 0 | 0 | 1 | 0
Not completed — Death | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | SPD476 (1.2 g) | SPD476 (2.4 g) | SPD476 (4.8 g) | Placebo | Total
Number analyzed (Participants) | 148 | 147 | 149 | 142 | 586
Age, Continuous [Mean (Standard Deviation); unit: years] — The Safety Population was used for this baseline measure. The Safety Population consists of subjects who were randomized and took at least 1 dose of investigational product. Out of the 592 subjects randomized, 6 were never dosed with investigational product. Therefore, 586 subjects are in the Safety Population.
  years | 57.8 (10.88) | 54.2 (10.10) | 56.7 (11.76) | 55.7 (11.15) | 56.1 (11.04)
Age, Customized [Count of Participants; unit: Participants] — The Safety Population was used for this baseline measure. The Safety Population consists of subjects who were randomized and took at least 1 dose of investigational product. Out of the 592 subjects randomized, 6 were never dosed with investigational product. Therefore, 586 subjects are in the Safety Population.
  Participants
    18 to < 35 years | 1 | 4 | 5 | 6 | 16
    35 to < 45 years | 16 | 21 | 18 | 16 | 71
    45 to < 55 years | 42 | 50 | 41 | 40 | 173
    55 to < 65 years | 45 | 48 | 45 | 45 | 183
    >= 65 years | 44 | 24 | 40 | 35 | 143
Sex: Female, Male [Count of Participants; unit: Participants] — The Safety Population was used for this baseline measure. The Safety Population consists of subjects who were randomized and took at least 1 dose of investigational product. Out of the 592 subjects randomized, 6 were never dosed with investigational product. Therefore, 586 subjects are in the Safety Population.
  Participants
    Female | 83 | 71 | 88 | 72 | 314
    Male | 65 | 76 | 61 | 70 | 272
Region of Enrollment [Count of Participants; unit: Participants] — This baseline measure consists of all randomized subjects (n = 592).
  Participants
    United States | 89 | 88 | 88 | 86 | 351
    Hungary | 2 | 3 | 6 | 3 | 14
    Canada | 5 | 5 | 4 | 5 | 19
    Finland | 4 | 5 | 5 | 4 | 18
    Brazil | 10 | 9 | 10 | 11 | 40
    Romania | 10 | 12 | 11 | 9 | 42
    South Africa | 14 | 16 | 15 | 15 | 60
    Netherlands | 5 | 3 | 5 | 5 | 18
    Germany | 7 | 6 | 4 | 4 | 21
    Italy | 2 | 1 | 2 | 4 | 9

OUTCOME MEASURES:

1. Primary Outcome: Percent of Subjects Without Recurrence of Diverticulitis
Description: Recurrence of diverticulitis is defined as the presence of each and all of the following 3 items: 1) abdominal pain, 2) a 15% increase in white blood cell count from baseline, 3) bowel wall thickening (>5 mm) and/or fat stranding as evidenced by spiral computerized axial tomography (CT) scan; OR surgical intervention for diverticular disease. Withdrawals are considered as recurrences.
Time Frame: up to 104 Weeks
Population: Full Analysis Set (FAS) consists of all subjects who were randomized and took at least 1 dose of investigational product.
Measure: Number; unit: percentage of subjects
Arm/Group | SPD476 (1.2 g) | SPD476 (2.4 g) | SPD476 (4.8 g) | Placebo
Number analyzed (Participants) | 148 | 147 | 149 | 142
percentage of subjects | 62.8 | 59.2 | 69.1 | 67.6
Statistical Analysis 1: Comparison: SPD476 (4.8 g) vs Placebo; Test type: Superiority or Other; p = 0.778, Cochran-Mantel-Haenszel
Statistical Analysis 2: Comparison: SPD476 (2.4 g) vs Placebo; Test type: Superiority or Other; p = 0.159, Cochran-Mantel-Haenszel
Statistical Analysis 3: Comparison: SPD476 (1.2 g) vs Placebo; Test type: Superiority or Other; p = 0.368, Cochran-Mantel-Haenszel

2. Secondary Outcome: Percent of Subjects Who Are CT-Recurrence Free of Diverticulitis
Description: CT-recurrence of diverticulitis is defined as: a positive spiral CT scan for diverticulitis showing, at a minimum, fat stranding with or without bowel wall thickening >5 mm or surgical intervention for diverticular disease. Withdrawals considered as CT-recurrences.
Time Frame: up to 104 weeks
Population: Full Analysis Set
Measure: Number; unit: percentage of subjects
Arm/Group | SPD476 (1.2 g) | SPD476 (2.4 g) | SPD476 (4.8 g) | Placebo
Number analyzed (Participants) | 148 | 147 | 149 | 142
percentage of subjects | 62.8 | 59.2 | 69.1 | 66.9
Statistical Analysis 1: Comparison: SPD476 (4.8 g) vs Placebo; Test type: Superiority or Other; p = 0.685, Cochran-Mantel-Haenszel
Statistical Analysis 2: Comparison: SPD476 (2.4 g) vs Placebo; Test type: Superiority or Other; p = 0.198, Cochran-Mantel-Haenszel
Statistical Analysis 3: Comparison: SPD476 (1.2 g) vs Placebo; Test type: Superiority or Other; p = 0.441, Cochran-Mantel-Haenszel

3. Secondary Outcome: Number of CT Scans Performed Within 7 Days of Suspected Recurrence of Diverticulitis That Were Positive
Description: A positive CT scan was defined as a CT scan that showed bowel wall thickening (>5 mm) and/or fat stranding as read by the central reader.
Time Frame: up to 104 Weeks
Population: Suspected Recurrence of Diverticulitis consists of subjects in the Full Analysis Set who had a CT scan performed. Since subjects may have had more than one suspected recurrence, counts are of the number of CT scans, not the number of subjects.
Measure: Number; unit: Number of CT Scans
Arm/Group | SPD476 (1.2 g) | SPD476 (2.4 g) | SPD476 (4.8 g) | Placebo
Number analyzed (Participants) | 55 | 52 | 51 | 40
Number of CT Scans
  Positive | 49 | 45 | 35 | 30
  Presence of abdominal pain | 48 | 39 | 34 | 29
  15% increase in WBC from baseline | 23 | 24 | 18 | 11
  Abdominal pain + 15% increase in WBC | 23 | 22 | 18 | 11

4. Secondary Outcome: Number of CT Scans Performed Within 7 Days of Suspected Recurrence of Diverticulitis That Were Negative
Description: A negative CT scan was defined as a CT scan that did not show bowel wall thickening (>5 mm) and/or fat stranding as read by the central reader.
Time Frame: up to 104 weeks
Population: as for outcome 3
Measure: Number; unit: Number of CT Scans
Arm/Group | SPD476 (1.2 g) | SPD476 (2.4 g) | SPD476 (4.8 g) | Placebo
Number analyzed (Participants) | 55 | 52 | 51 | 40
Number of CT Scans
  Negative | 9 | 8 | 22 | 15
  Presence of abdominal pain | 8 | 6 | 17 | 12
  15% increase in WBC from Baseline | 1 | 2 | 4 | 4
  Abdominal pain + 15% increase in WBC | 1 | 2 | 4 | 3

5. Secondary Outcome: Number of CT Scans Performed More Than 7 Days From Suspected Recurrence of Diverticulitis That Were Positive
Description: as for outcome 3
Time Frame: up to 104 weeks
Population: as for outcome 3
Measure: Number; unit: Number of CT Scans
Arm/Group | SPD476 (1.2 g) | SPD476 (2.4 g) | SPD476 (4.8 g) | Placebo
Number analyzed (Participants) | 55 | 52 | 51 | 40
Number of CT Scans
  Positive | 0 | 0 | 1 | 1
  Presence of abdominal pain | 0 | 0 | 0 | 1
  15% increase in WBC from baseline | 0 | 0 | 0 | 0
  Abdominal pain + 15% increase in WBC | 0 | 0 | 0 | 0

6. Secondary Outcome: Number of CT Scans Performed More Than 7 Days From Suspected Recurrence of Diverticulitis That Were Negative
Description: as for outcome 4
Time Frame: up to 104 weeks
Population: as for outcome 3
Measure: Number; unit: Number of CT Scans
Arm/Group | SPD476 (1.2 g) | SPD476 (2.4 g) | SPD476 (4.8 g) | Placebo
Number analyzed (Participants) | 55 | 52 | 51 | 40
Number of CT Scans
  Negative | 1 | 0 | 0 | 0
  Presence of abdominal pain | 1 | 0 | 0 | 0
  15% increase in WBC from baseline | 0 | 0 | 0 | 0
  Abdominal pain + 15% increase in WBC | 0 | 0 | 0 | 0

7. Secondary Outcome: Percent of Subjects Requiring Surgery for Diverticulitis
Time Frame: up to 104 Weeks
Population: Full Analysis Set
Measure: Number; unit: percentage of subjects
Arm/Group | SPD476 (1.2 g) | SPD476 (2.4 g) | SPD476 (4.8 g) | Placebo
Number analyzed (Participants) | 148 | 147 | 149 | 142
percentage of subjects | 4.7 | 2.7 | 2.0 | 1.4

ADVERSE EVENTS:
Arm/Group | SPD476 (1.2 g) | SPD476 (2.4 g) | SPD476 (4.8 g) | Placebo
Serious Adverse Events (participants affected / at risk) | 9/148 | 13/147 | 14/149 | 15/142
Other Adverse Events (participants affected / at risk) | 108/148 | 111/147 | 110/149 | 105/142
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | SPD476 (1.2 g) (N=148) | SPD476 (2.4 g) (N=147) | SPD476 (4.8 g) (N=149) | Placebo (N=142)
Agranulocytosis (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Angina pectoris (Cardiac disorders) | 0 | 1 | 1 | 1
Atrial fibrillation (Cardiac disorders) | 1 | 1 | 0 | 0
Cardiac failure (Cardiac disorders) | 0 | 0 | 1 | 0
Ventricular extrasystoles (Cardiac disorders) | 0 | 1 | 0 | 0
Supraventricular tachycardia (Cardiac disorders) | 1 | 0 | 0 | 0
Gastroesophogeal reflux disease (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Small intestinal hemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Hiatus hernia (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Esophagitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Abdominal pain lower (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Mallory-Weiss syndrome (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Chest pain (General disorders) | 0 | 0 | 2 | 0
Multi-organ failure/Death (General disorders) | 0 | 1 | 0 | 0
Chest discomfort (General disorders) | 1 | 0 | 0 | 0
Cholangitis acute (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 1 | 0 | 1 | 2
Subcutaneous abscess (Infections and infestations) | 0 | 0 | 1 | 0
Appendicitis (Infections and infestations) | 0 | 1 | 0 | 0
Bronchitis (Infections and infestations) | 1 | 0 | 0 | 0
Peridiverticular abscess (Infections and infestations) | 1 | 0 | 0 | 0
Pharyngitis (Infections and infestations) | 1 | 0 | 0 | 0
Borrelia infection (Infections and infestations) | 0 | 0 | 0 | 1
Pneumonia viral (Infections and infestations) | 0 | 0 | 0 | 1
Viral pericarditis (Infections and infestations) | 0 | 0 | 0 | 1
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Patella fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Post procedural edema (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Radius fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Hip fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Ovarian granulosa-theca cell tumor (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Cardiac neoplasm unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 0 | 2 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 1 | 0
Transient ischemic attack (Nervous system disorders) | 1 | 0 | 0 | 0
Panic attack (Psychiatric disorders) | 0 | 0 | 0 | 1
Ovarian cyst (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
Uterovaginal prolapse (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1
Hypotension (Vascular disorders) | 0 | 1 | 0 | 0
Intra-abdominal hemorrhage (Vascular disorders) | 0 | 1 | 0 | 0
Femoral arterial stenosis (Vascular disorders) | 0 | 0 | 0 | 1
Hemorrhage (Vascular disorders) | 0 | 0 | 0 | 1
Hypertension (Vascular disorders) | 0 | 0 | 0 | 1
Thrombosis (Vascular disorders) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | SPD476 (1.2 g) (N=148) | SPD476 (2.4 g) (N=147) | SPD476 (4.8 g) (N=149) | Placebo (N=142)
Abdominal pain (Gastrointestinal disorders) | 19 | 19 | 15 | 12
Diarrhea (Gastrointestinal disorders) | 15 | 15 | 18 | 12
Nausea (Gastrointestinal disorders) | 5 | 8 | 10 | 11
Dyspepsia (Gastrointestinal disorders) | 5 | 11 | 6 | 6
Constipation (Gastrointestinal disorders) | 9 | 6 | 6 | 12
Abdominal pain lower (Gastrointestinal disorders) | 5 | 2 | 10 | 7
Urinary tract infection (Infections and infestations) | 11 | 14 | 10 | 7
Sinusitis (Infections and infestations) | 12 | 8 | 10 | 11
Influenza (Infections and infestations) | 11 | 8 | 9 | 11
Bronchitis (Infections and infestations) | 8 | 7 | 9 | 7
Nasopharyngitis (Infections and infestations) | 5 | 10 | 8 | 9
Back pain (Musculoskeletal and connective tissue disorders) | 10 | 11 | 11 | 12
Headache (Nervous system disorders) | 14 | 10 | 14 | 13
Cough (Respiratory, thoracic and mediastinal disorders) | 9 | 3 | 4 | 2
Hypertension (Vascular disorders) | 6 | 8 | 2 | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If a multicenter publication is not submitted within twelve (12) months after conclusion, abandonment or termination of the Study at all sites, or after Sponsor confirms there shall be no multicenter Study publication, the Institution and/or such Principal Investigator may publish the results from the Institution site individually.